CLINICAL TRIAL: NCT00918502
Title: Adherent Respiratory Monitoring for Apnea Detection and Evaluation Study
Brief Title: Monitor Patients With Sleep Apnea
Acronym: ARMADA
Status: Completed | Type: Observational
Sponsor: Corventis, Inc. (Industry)
Responsible Party: Madhuri Bhat, VP Regulatory and Clinical affairs, Corventis
Other Study IDs: COR-2009-004
Record Dates: First submitted 2009-06-10; First posted 2009-06-11 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2010-02

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: AVIVO system — Non invasive external monitoring device

SUMMARY:
The primary objective of the study is to gather data to correlate physiological signals measured by the AVIVO™ Mobile Patient Management System with the patient's respiratory status, including apnea and hypopnea events, during polysomnography

DETAILED DESCRIPTION:
Patients with suspected sleep disordered breathing will be monitored during polysomnography and the collected information will be used to assess patient's respiratory status.

ELIGIBILITY:
Inclusion Criteria:

* Is female or male, 18 years of age or older
* Undergoing polysomnography for suspected sleep apnea
* Is willing to provide written informed consent and comply with study guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: sleep study
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Imad Libbus, PhD, Study Director — Corventis, Inc.